CLINICAL TRIAL: NCT07085078
Title: Effects of Progressive Relaxation Exercise on Menopausal Symptoms and Work Performance: A Randomized Control Study
Brief Title: Progressive Relaxation Exercise, Menopausal Symptoms and Working Performance
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Collaborators: Uludag University (Other)
Responsible Party: Principal Investigator, Gonca Buran, Assoc. Prof., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18/17
Record Dates: First submitted 2025-06-26; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Menopause; Menopause Related Conditions
Keywords: menophose; work performance; progressive relaxation; menopausal symptoms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): Progressive relaxation exercis
  Interventions: Behavioral: progressive relaxation exercises
- Control (No Intervention): Participants with menopausal symptoms assigned to the control group will not receive any intervention. They are expected to answer the scale questions used in the study.

INTERVENTIONS:
Behavioral: progressive relaxation exercises — Participants with menopausal symptoms received progressive relaxation exercise training, led by the responsible researcher who assigned them to the experimental group.
  Arms: Education

SUMMARY:
Women typically enter menopause between the ages of 40 and 47, and they spend approximately one-third of their lives in this phase. During menopause, many experience hot flashes due to decreased estrogen levels, along with vasomotor changes such as altered heart rhythms and sleep disturbances. These issues may accompany or occur independently of hot flashes. Additionally, psychological changes can arise, including tension, sudden mood swings, anxiety, stress, and depression. Physiological concerns may include vaginal atrophy and stress incontinence.

DETAILED DESCRIPTION:
Previous studies have shown that menopausal symptoms can significantly increase women's social appearance anxiety, depression, stress, and anxiety overall, negatively impacting their quality of life. Moreover, a limited number of recent studies have attempted to explore the relationship between the severity of menopausal symptoms in the workplace and factors such as job performance, career development decisions, and overall work participation.

This study aims to investigate the effects of progressive relaxation exercises on women's menopausal symptoms and their work performance.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman between the ages of 45-65
* Being able to read and understand Turkish
* Being at least a primary school graduate
* Not having menstruation for a year

Exclusion Criteria:

* Having a disability in maintaining communication (such as hearing and speaking)
* Having entered early menopause (no menstruation) through surgery or natural means,
* Being on hormone therapy
* Filling out forms incompletely

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants are eligible as menopausal symptoms will be assessed
Enrollment: 106 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Personal information form before intervention | Day 1 (During recruitment)
  Evaluation of women using personal information.
  This tool includes questions on women's sociodemographic characteristics
Before intervention, menopausal symptoms | Day 1 (during recruitment)
  Evaluation of menopausal symptoms with Menopause Rating Scale (MRS). It is a Likert-type scale consisting of 11 items, including menopausal complaints. For each item, there are options of "0= None", "1= Mild", "2= Moderate", "3= Severe", and "4= Very severe". The lowest possible score is 0, the highest score is 44. An increase in the total score obtained from the scale indicates an increase in the severity of the complaints experienced.
Before intervention, Individual work performance | Day 1 (During recruitment)
  Before intervention, participants are evaluated with the "Individual Work Performance Questionnaire"The scale was designed to measure job performance perception. It consists of 18 Likert-type items. A high score on the scale indicates that job performance perception has increased.

SECONDARY OUTCOMES:
After intervention, menopausal symptoms | Ten days after the conclusion of the five-week training program.
  Evaluation of menopausal symptoms with Menopause Rating Scale (MRS). (The lowest possible score is 0, the highest score is 44. The increase in the total score obtained from the scale indicates an increase in the severity of the complaints).
After intervention, Individual work performance | Ten days after the conclusion of the five-week training program.
  participants are evaluated with the "Individual Work Performance Questionnaire" (The scale was designed to measure job performance perception. It consists of 18 Likert-type items. A high score on the scale indicates that job performance perception has increased.)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bursa Uludağ Üniversitesi, Nilufer, Bursa
  - Bursa Uludag University, Bursa

IPD SHARING:
Plan to Share IPD: Yes
The responsible researcher will apply the training and exercises and code the data as A and B. A and B will be coded as A and B. The second researcher will apply the question and scale forms coded as A and B. The third researcher will not know which group the A and B data belong to, and the data will be entered into the SPSS program as A and B groups. The analyses will be carried out by the researcher who is blind to the groups. After the analyses are completed, all researchers will know which arm the findings belong to A and B groups. They will be able to access all of the data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: I have a plan to make IPD available. A data dictionary (a description of the variables or types of data collected for each individual) will be provided so that the data can be fully interpreted.
Access Criteria: IPD and information will be accessible to researchers and institutional auditors who are assisting with the information. The types of analyses and methods for these analyses that are appropriate for data sharing do not need to be approved by independent review.
URL: https://tip.uludag.edu.tr/arastirma/bap

REFERENCES:
- [Result] O'Neill MT, Jones V, Reid A. Impact of menopausal symptoms on work and careers: a cross-sectional study. Occup Med (Lond). 2023 Sep 29;73(6):332-338. doi: 10.1093/occmed/kqad078. PMID 37542726
- [Result] Koopmans L, Bernaards CM, Hildebrandt VH, Lerner D, de Vet HC, van der Beek AJ. Cross-cultural adaptation of the Individual Work Performance Questionnaire. Work. 2015;53(3):609-19. doi: 10.3233/WOR-152237. PMID 26835864